CLINICAL TRIAL: NCT05452447
Title: A Cluster Randomized, Placebo Control Trial to Evaluate the Efficacy of a Spatial Repellent (Mosquito ShieldTM) Against Aedes-borne Virus Infection Among Children ≥ 4-16 Years of Age in the Gampaha District, Sri Lanka
Brief Title: Spatial Repellents for Aedes-borne Virus Control in Sri Lanka
Acronym: AEGIS ABV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: S.C. Johnson & Son, Inc. (Industry); fhiClinical (Unknown); Ministry of Health, Sri Lanka (Other Government); University of Sri Jayewardenepura, Sri Lanka (Unknown); University of Washington (Other); RemediumOne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-05-6629
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Arbovirus Infections
Keywords: Dengue; Zika; Chikungunya; Spatial Repellent; Transfluthrin; Vector-borne diseases; Mosquito vectors; Incidence
MeSH Terms: conditions — Arbovirus Infections; Dengue; Zika Virus Infection; Chikungunya Fever; Vector Borne Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spatial Repellent (Experimental): Transfluthrin
  Interventions: Device: Transfluthrin
- Placebo (Placebo Comparator): Inert ingredients
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transfluthrin — Passive emanator with formulated transfluthrin
  Arms: Spatial Repellent
Device: Placebo — Passive emanator with formulated inert ingredients
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate and quantify the protective efficacy (PE) of a single SR product, in reducing DENV infection and active Aedes-borne virus (ABV) disease in human cohorts. The study design will be a prospective, cluster randomized controlled trial (cRCT). Although not a specific objective of this project, an overall goal is to allow for official recommendations (or not) from the World Health Organization (WHO) for the use of SRs in public health. A WHO global policy recommendation will establish evaluation systems of SR products to regulate efficacy evaluations, thereby increasing quality, overall use and a consequent reduction in disease.

DETAILED DESCRIPTION:
The study will be a prospective, cRCT, participant and observer-blinded, placebo-controlled trial in a site endemic for ABV to measure the impact of a SR product on new ABV virus infections. Clusters of households, each cluster containing 110-120 residents testing negative for antibodies against DENV (seronegative) or positive to a single DENV infection (monotypic), will be selected from three MOH areas in the district of Gampaha: Negambo, Wattala, Kelaniya. All participating houses in each cluster will be monitored entomologically for adult Aedes aegypti surveys for 3 months before deployment of the SR intervention and monthly after the intervention is in place. Entomological surveys will include monitoring of indoor Ae. aegypti adult population densities and blood-fed status. DENV infection in study participants will be assessed by serologic testing of scheduled longitudinal blood samples (primary outcome) and passively by monitoring febrile persons for acute Dengue illness (secondary outcome). Seroconversion to DENV from baseline (pre-intervention) and follow-up (post-intervention) samples as well as ABV active disease rates will be compared between active intervention and placebo (control) clusters. Testing and confirmation of Zika virus (ZIKV) and Chikungunya virus (CHIKV) infection at baseline and during the intervention phase of the trial will be dependent on circulation history/detection in study area during study period.

The spatial repellent (SR) will be a new formulation of transfluthrin. This active ingredient (AI) is widely used in mosquito coils and other household pest control products worldwide. The new formulation is a passive emanator that will release the AI over a period of up to four weeks, Mosquito ShieldTM. The emanator will consist of a pre-treated piece of cellulose acetate or other medium, which will be positioned within consenting households according to manufacturer specifications of 2 units/9m2. A placebo product of matched design with inert ingredients will be applied similarly. The Mosquito ShieldTM and placebo products for this study will be designed and provided by S.C. Johnson, INC. A Family Company.

ELIGIBILITY:
LONGITUDINAL SEROCONVERSION Individual Level

Inclusion Criteria:

* ≥ 4 - 16 years of age
* Plans to stay in residence and/or study area for a minimum of 24 months
* Resident of household or frequent visitor (~20% of day hours in house / month)

Exclusion Criteria:

* < 4 and > 16 years of age
* Plans to leave residence and/or study area within next 24 months
* Temporary visitor to household (<20% of day hours in house/ month)

FEBRILE SURVEILLANCE Household Level

Inclusion Criteria:

* Adult head of households agrees to census, health visits and logging resident symptoms when febrile (or in the case of suspected Zika in the absence of fever, presenting with rash, arthralgia, arthritis or non-purulent conjunctivitis).
* Individuals spend a minimum of 4hrs per week during the daytime hours or sleep in the house.

Exclusion Criteria:

* Adult head of households does not agree to census, health visits or logging symptoms of residents.
* Households where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).
* Sites where no residents spend time during the day (i.e. work 7d a week outside the home).

FEBRILE SURVEILLANCE Individual Level

Inclusion Criteria:

* ≥ 6mo of age.
* Fever at the time of presentation or report of feverishness within the previous 24 hours or presenting with a rash, arthralgia, arthritis or non-purulent conjunctivitis (suspicion of ZIKA determined by project physician)
* Individual who spends a minimum of 4 hours per week within the household or sleeps in the house.

Exclusion Criteria:

* < 6mo of age.
* No fever at time of presentation or report of feverishness within the previous 24 hours or not reporting with a rash, arthralgia, arthritis or non-purulent conjunctivitis
* Individuals who have spent less than 4 hours in the household during the week prior to illness.

ENTOMOLOGICAL MONITORING Household Level

Inclusion Criteria:

* Adult head of household agrees to surveys.
* Properties where study personnel do not identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).

Exclusion Criteria:

* Adult head of household does not agree to surveys.
* Properties where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).

SPATIAL REPELLENT INTERVENTION Household Level

Inclusion Criteria:

* Adult head of households agrees to have intervention applied inside the home and to provide access to team member at 4-week intervals to change products.
* Properties where study personnel do not identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).

Exclusion Criteria:

* Adult head of household does not agree to Mosquito ShieldTM deployment or study team access.
* Properties where study personnel identify a security risk (i.e., site where drugs are sold, residents are always drunk or hostile).

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6949 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Aedes-borne virus (ABV) infection in the 'longitudinal cohort'. | 24 months
  The primary endpoint is the fraction of monotypic or seronegative individuals in the 'longitudinal cohort' who seroconvert to an arbovirus during the follow-up period post randomization with intervention. Here, the intervention follow-up period is 2 years after initial deployment of SR or placebo. There will be 3 blood samplings from longitudinal cohort participants for measure of seroconversion: one for baseline serostatus characterization (T0), a second at 12 months (T1) and a third at 24 months (T2) from time of initial placement of intervention.

SECONDARY OUTCOMES:
Clinically apparent cases of Aedes-borne virus (ABV) disease. | 24 months
  Clinically apparent is defined as an acute infection that causes overt symptoms (fever, rash, etc.) indicating virus circulation in the blood. For the longitudinal cohort participants, acute and convalescent blood sampling based on time of health facility visit when febrile throughout the intervention period. For other household members participating in febrile surveillance, case definition measured and reported whenever they visit designated health facilities throughout the intervention period.
Adult female Aedes aegypti indoor abundance. | 24 months
  Measured by comparing adult female Aedes aegypti indoor abundance in households using Procopak mosquito aspiration with active and placebo product receiving standard entomological surveillance and control procedures by the local Ministry of Health, as an indicator for reduced mosquito house entry due to effect of product. Indoor mosquito collections in enrolled households once every 28 days during intervention.
Adult female Aedes aegypti blood fed rate. | 24 months
  Measured by comparing adult female Aedes aegypti blood fed rate in households with active and placebo product receiving standard entomological surveillance and control procedures by the local Ministry of Health, as an indicator for reduced mosquito human contact due to effect of product. Direct mosquito abdominal observation by microscopy from samples taken by Procopak aspiration during indoor mosquito collections in enrolled households once every 28 days during intervention.
Diversion of Aedes aegypti mosquitoes into untreated houses. | 24 months
  Measured by comparing adult female Aedes aegypti abundance using Procopak mosquito aspiration in untreated households adjacent to treatment clusters (with active product) to untreated households adjacent to placebo clusters as an indicator for mosquito diversion due to effect of product. Indoor mosquito collections in enrolled households once every 28 days during intervention.
Overall incidence of Aedes-borne virus (ABV) infection. | 24 months
  Measured by the seroconversion rates of all children enrolled in the trial, independent of order of infection (i.e., including tertiary and quaternary infections). Based on blood samples taken for longitudinal seroconversion and febrile surveillance from time of initial placement of intervention.

OTHER OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs). | 24 months
  Measured by solicited and unsolicited reports from both the longitudinal cohort and febrile surveillance cohort during the trial period. Mean, minimum and maximum frequency and percentage of AEs and SAEs across clusters among enrolled subjects will be summarized by treatment arm.
Incidence of Aedes-borne virus (ABV) infection in subjects residing in households within treatment clusters but without SR product. | 24 months
  Measured by comparing Aedes-borne virus infection rates between subjects residing in households with SR product in treatment clusters and subjects from the same clusters who did not agree to the SR application in their households but are receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator of community effect due to effect of product.
Clinically apparent cases of Aedes-borne virus (ABV) disease in subjects residing in households within treatment clusters but without SR product. | 24 months
  Measured by comparing Aedes-borne virus disease case rates between subjects residing in households with SR product in households in treatment clusters and individuals from the same clusters who did not agree to the SR application in their households but are receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator of community effect due to effect of product.
Adult female Aedes aegypti indoor abundance using Procopak mosquito aspiration in households within treatment clusters but without SR product. | 24 months
  Measured by comparing adult female Aedes aegypti indoor abundance in households with SR product in treatment clusters and households from the same clusters who did not agree to the SR application but are receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator of community effect to effect of product. Indoor mosquito collections in enrolled households once every 28 days during intervention
Adult female Aedes aegypti blood fed rate using Procopak mosquito aspiration in households within treatment clusters but without SR product. | 24 months
  Measured by comparing adult female Aedes aegypti blood fed rate in households with SR product in treatment clusters and households from the same clusters who did not agree to the SR application but are receiving standard entomological surveillance and control procedures by the local ministry of health, as an indicator of community effect to effect of product. Samples from indoor mosquito collections in enrolled households once every 28 days during intervention.

CONTACTS AND LOCATIONS:
Overall Officials: John P Grieco, Ph.D., Study Director — University of Notre Dame; Korelege Hasitha Aravinda Tissera, M.D., Principal Investigator — Epidemiology Unit, Ministry of Health, Sri Lanka
Locations (2):
- Sri Lanka (2):
  - Epidemiology Unit, Ministry of Health, Colombo, West
  - Clinical Trials Unit, Ragama, West

IPD SHARING:
Plan to Share IPD: Yes
Analytical datasets will be anonymized and GPS tag-blurred to remove sensitive information prior to sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data and supporting information will be made available 12 months following completion of data analysis and will remain open access in the public domain.
Access Criteria: Open-access repository distributed under the terms of the Creative Commons Attribution (CC-BY) License, which permits unrestricted use, distribution, and reproduction in any medium, provided the original author and source are credited.

REFERENCES:
- [Background] Achee NL, Bangs MJ, Farlow R, Killeen GF, Lindsay S, Logan JG, Moore SJ, Rowland M, Sweeney K, Torr SJ, Zwiebel LJ, Grieco JP. Spatial repellents: from discovery and development to evidence-based validation. Malar J. 2012 May 14;11:164. doi: 10.1186/1475-2875-11-164. PMID 22583679
- [Background] Achee NL, Sardelis MR, Dusfour I, Chauhan KR, Grieco JP. Characterization of spatial repellent, contact irritant, and toxicant chemical actions of standard vector control compounds. J Am Mosq Control Assoc. 2009 Jun;25(2):156-67. doi: 10.2987/08-5831.1. PMID 19653497
- [Background] Ansari MZ, Shope RE, Malik S. Evaluation of vero cell lysate antigen for the ELISA of flaviviruses. J Clin Lab Anal. 1993;7(4):230-7. doi: 10.1002/jcla.1860070408. PMID 8395596
- [Background] Comach G, Blair PJ, Sierra G, Guzman D, Soler M, de Quintana MC, Bracho-Labadie M, Camacho D, Russell KL, Olson JG, Kochel TJ. Dengue virus infections in a cohort of schoolchildren from Maracay, Venezuela: a 2-year prospective study. Vector Borne Zoonotic Dis. 2009 Feb;9(1):87-92. doi: 10.1089/vbz.2007.0213. Epub 2008 Sep 12. PMID 18788903
- [Background] Forshey BM, Morrison AC, Cruz C, Rocha C, Vilcarromero S, Guevara C, Camacho DE, Alava A, Madrid C, Beingolea L, Suarez V, Comach G, Kochel TJ. Dengue virus serotype 4, northeastern Peru, 2008. Emerg Infect Dis. 2009 Nov;15(11):1815-8. doi: 10.3201/eid1511.090663. PMID 19891873
- [Background] Erlanger TE, Keiser J, Utzinger J. Effect of dengue vector control interventions on entomological parameters in developing countries: a systematic review and meta-analysis. Med Vet Entomol. 2008 Sep;22(3):203-21. doi: 10.1111/j.1365-2915.2008.00740.x. PMID 18816269
- [Background] Getis A, Morrison AC, Gray K, Scott TW. Characteristics of the spatial pattern of the dengue vector, Aedes aegypti, in Iquitos, Peru. Am J Trop Med Hyg. 2003 Nov;69(5):494-505. PMID 14695086
- [Background] Grieco JP, Achee NL, Chareonviriyaphap T, Suwonkerd W, Chauhan K, Sardelis MR, Roberts DR. A new classification system for the actions of IRS chemicals traditionally used for malaria control. PLoS One. 2007 Aug 8;2(8):e716. doi: 10.1371/journal.pone.0000716. PMID 17684562
- [Background] Grieco JP, Achee NL, Sardelis MR, Chauhan KR, Roberts DR. A novel high-throughput screening system to evaluate the behavioral response of adult mosquitoes to chemicals. J Am Mosq Control Assoc. 2005 Dec;21(4):404-11. doi: 10.2987/8756-971X(2006)21[404:ANHSST]2.0.CO;2. PMID 16506566
- [Background] Grieco JP, Achee NL, Andre RG, Roberts DR. A comparison study of house entering and exiting behavior of Anopheles vestitipennis (Diptera: Culicidae) using experimental huts sprayed with DDT or deltamethrin in the southern district of Toledo, Belize, C.A. J Vector Ecol. 2000 Jun;25(1):62-73. PMID 10925798
- [Background] Gubler DJ. Aedes aegypti and Aedes aegypti-borne disease control in the 1990s: top down or bottom up. Charles Franklin Craig Lecture. Am J Trop Med Hyg. 1989 Jun;40(6):571-8. doi: 10.4269/ajtmh.1989.40.571. No abstract available. PMID 2472746
- [Background] Gubler DJ. Dengue and dengue hemorrhagic fever. Clin Microbiol Rev. 1998 Jul;11(3):480-96. doi: 10.1128/CMR.11.3.480. PMID 9665979
- [Background] Gubler DJ. Epidemic dengue/dengue hemorrhagic fever as a public health, social and economic problem in the 21st century. Trends Microbiol. 2002 Feb;10(2):100-3. doi: 10.1016/s0966-842x(01)02288-0. PMID 11827812
- [Background] Hapuarachchi HA, Bandara KB, Hapugoda MD, Williams S, Abeyewickreme W. Laboratory confirmation of dengue and chikungunya co-infection. Ceylon Med J. 2008 Sep;53(3):104-5. doi: 10.4038/cmj.v53i3.252. No abstract available. PMID 18982804
- [Background] Hapuarachchi HC, Bandara KB, Sumanadasa SD, Hapugoda MD, Lai YL, Lee KS, Tan LK, Lin RT, Ng LF, Bucht G, Abeyewickreme W, Ng LC. Re-emergence of Chikungunya virus in South-east Asia: virological evidence from Sri Lanka and Singapore. J Gen Virol. 2010 Apr;91(Pt 4):1067-76. doi: 10.1099/vir.0.015743-0. Epub 2009 Dec 2. PMID 19955565
- [Background] Hayes CG, Phillips IA, Callahan JD, Griebenow WF, Hyams KC, Wu SJ, Watts DM. The epidemiology of dengue virus infection among urban, jungle, and rural populations in the Amazon region of Peru. Am J Trop Med Hyg. 1996 Oct;55(4):459-63. doi: 10.4269/ajtmh.1996.55.459. PMID 8916809
- [Background] Innis BL, Nisalak A, Nimmannitya S, Kusalerdchariya S, Chongswasdi V, Suntayakorn S, Puttisri P, Hoke CH. An enzyme-linked immunosorbent assay to characterize dengue infections where dengue and Japanese encephalitis co-circulate. Am J Trop Med Hyg. 1989 Apr;40(4):418-27. doi: 10.4269/ajtmh.1989.40.418. PMID 2540664
- [Background] Kanakaratne N, Wahala WM, Messer WB, Tissera HA, Shahani A, Abeysinghe N, de-Silva AM, Gunasekera M. Severe dengue epidemics in Sri Lanka, 2003-2006. Emerg Infect Dis. 2009 Feb;15(2):192-9. doi: 10.3201/eid1502.080926. PMID 19193262
- [Background] Kawada H, Maekawa Y, Tsuda Y, Takagi M. Laboratory and field evaluation of spatial repellency with metofluthrin-impregnated paper strip against mosquitoes in Lombok Island, Indonesia. J Am Mosq Control Assoc. 2004 Sep;20(3):292-8. PMID 15532930
- [Background] Kawada H, Maekawa Y, Tsuda Y, Takagi M. Trial of spatial repellency of metofluthrin-impregnated paper strip against Anopheles and Culex in shelters without walls in Lombok, Indonesia. J Am Mosq Control Assoc. 2004 Dec;20(4):434-7. PMID 15669387
- [Background] Kawada H, Maekawa Y, Takagi M. Field trial on the spatial repellency of metofluthrin-impregnated plastic strips for mosquitoes in shelters without walls (beruga) in Lombok, Indonesia. J Vector Ecol. 2005 Dec;30(2):181-5. PMID 16599150
- [Background] Kochel TJ, Watts DM, Halstead SB, Hayes CG, Espinoza A, Felices V, Caceda R, Bautista CT, Montoya Y, Douglas S, Russell KL. Effect of dengue-1 antibodies on American dengue-2 viral infection and dengue haemorrhagic fever. Lancet. 2002 Jul 27;360(9329):310-2. doi: 10.1016/S0140-6736(02)09522-3. PMID 12147378
- [Background] Kularatne SA, Gihan MC, Weerasinghe SC, Gunasena S. Concurrent outbreaks of Chikungunya and Dengue fever in Kandy, Sri Lanka, 2006-07: a comparative analysis of clinical and laboratory features. Postgrad Med J. 2009 Jul;85(1005):342-6. doi: 10.1136/pgmj.2007.066746. PMID 19581242
- [Background] Kuno G. Review of the factors modulating dengue transmission. Epidemiol Rev. 1995;17(2):321-35. doi: 10.1093/oxfordjournals.epirev.a036196. No abstract available. PMID 8654514
- [Background] Lanciotti RS, Calisher CH, Gubler DJ, Chang GJ, Vorndam AV. Rapid detection and typing of dengue viruses from clinical samples by using reverse transcriptase-polymerase chain reaction. J Clin Microbiol. 1992 Mar;30(3):545-51. doi: 10.1128/jcm.30.3.545-551.1992. PMID 1372617
- [Background] Lucas JR, Shono Y, Iwasaki T, Ishiwatari T, Spero N, Benzon G. U.S. laboratory and field trials of metofluthrin (SumiOne) emanators for reducing mosquito biting outdoors. J Am Mosq Control Assoc. 2007 Mar;23(1):47-54. doi: 10.2987/8756-971X(2007)23[47:ULAFTO]2.0.CO;2. PMID 17536367
- [Background] Messer WB, Vitarana UT, Sivananthan K, Elvtigala J, Preethimala LD, Ramesh R, Withana N, Gubler DJ, De Silva AM. Epidemiology of dengue in Sri Lanka before and after the emergence of epidemic dengue hemorrhagic fever. Am J Trop Med Hyg. 2002 Jun;66(6):765-73. doi: 10.4269/ajtmh.2002.66.765. PMID 12224589
- [Background] Monath TP. Dengue: the risk to developed and developing countries. Proc Natl Acad Sci U S A. 1994 Mar 29;91(7):2395-400. doi: 10.1073/pnas.91.7.2395. PMID 8146129
- [Background] Morens DM, Halstead SB, Repik PM, Putvatana R, Raybourne N. Simplified plaque reduction neutralization assay for dengue viruses by semimicro methods in BHK-21 cells: comparison of the BHK suspension test with standard plaque reduction neutralization. J Clin Microbiol. 1985 Aug;22(2):250-4. doi: 10.1128/jcm.22.2.250-254.1985. PMID 4031038
- [Background] Morrison AC, Minnick SL, Rocha C, Forshey BM, Stoddard ST, Getis A, Focks DA, Russell KL, Olson JG, Blair PJ, Watts DM, Sihuincha M, Scott TW, Kochel TJ. Epidemiology of dengue virus in Iquitos, Peru 1999 to 2005: interepidemic and epidemic patterns of transmission. PLoS Negl Trop Dis. 2010 May 4;4(5):e670. doi: 10.1371/journal.pntd.0000670. PMID 20454609
- [Background] Morrison AC, Zielinski-Gutierrez E, Scott TW, Rosenberg R. Defining challenges and proposing solutions for control of the virus vector Aedes aegypti. PLoS Med. 2008 Mar 18;5(3):e68. doi: 10.1371/journal.pmed.0050068. PMID 18351798
- [Background] Morrison AC, Astete H, Chapilliquen F, Ramirez-Prada C, Diaz G, Getis A, Gray K, Scott TW. Evaluation of a sampling methodology for rapid assessment of Aedes aegypti infestation levels in Iquitos, Peru. J Med Entomol. 2004 May;41(3):502-10. doi: 10.1603/0022-2585-41.3.502. PMID 15185957
- [Background] Morrison AC, Gray K, Getis A, Astete H, Sihuincha M, Focks D, Watts D, Stancil JD, Olson JG, Blair P, Scott TW. Temporal and geographic patterns of Aedes aegypti (Diptera: Culicidae) production in Iquitos, Peru. J Med Entomol. 2004 Nov;41(6):1123-42. doi: 10.1603/0022-2585-41.6.1123. PMID 15605653
- [Background] Munasinghe DR, Amarasekera PJ, Fernando CF. An epidemic of dengue-like fever in Ceylon (chikungunya--a clinical and haematological study. Ceylon Med J. 1966 Dec;11(4):129-42. No abstract available. PMID 5984948
- [Background] Ogoma SB, Moore SJ, Maia MF. A systematic review of mosquito coils and passive emanators: defining recommendations for spatial repellency testing methodologies. Parasit Vectors. 2012 Dec 7;5:287. doi: 10.1186/1756-3305-5-287. PMID 23216844
- [Background] Syafruddin D, Bangs MJ, Sidik D, Elyazar I, Asih PB, Chan K, Nurleila S, Nixon C, Hendarto J, Wahid I, Ishak H, Bogh C, Grieco JP, Achee NL, Baird JK. Impact of a spatial repellent on malaria incidence in two villages in Sumba, Indonesia. Am J Trop Med Hyg. 2014 Dec;91(6):1079-87. doi: 10.4269/ajtmh.13-0735. Epub 2014 Oct 13. PMID 25311699